CLINICAL TRIAL: NCT05370066
Title: Anonymized Data Collection From the CS6BP and Other Modalities for the Purpose of Developing Continuous, Absolute, Non-Inflating Measurement of Blood Pressure
Brief Title: Anonymized Data Collection From the CS6BP and Other Modalities for the Purpose Measurement of Blood Pressure
Acronym: BPW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CardiacSense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 007_BPW_DC_OS_BP; CL00600 (Registry Identifier: MOH)
Record Dates: First submitted 2022-04-18; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Blood Pressure

STUDY DESIGN:
Intervention Model Description: Data collection for algorithm development CS6BP data will be collected in parallel with commercially available blood pressure monitor measurement.
Masking Description: open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS6BP and cuff (Experimental): CS6BP watches will be used in the study with Commercially available FDA approved Blood pressure monitors:
  Interventions: Device: CS6BP watches will be used in the study.

INTERVENTIONS:
Device: CS6BP watches will be used in the study. — CS6BP watches will be used with FDA approved Blood pressure monitors
  Other Names: Comparator: Commercially available FDA approved Blood pressure monitors

SUMMARY:
This study is performed on hospitalized subjects in the Internal Medicine Division. The study is intended for data collection. The data will be obtained from commercially available blood pressure monitors and simultaneously from the CS6BP watch.

DETAILED DESCRIPTION:
This is a prospective open-label study. Hospitalized subjects from Internal Medicine Division will be measured simultaneously with a commercially available blood pressure monitor and CS6BP watch. Subjects may be measured at the clinic or home up to one month following their discharge from the hospital.

Screening:

PI or delegated physician will confirm the eligibility of subjects. Eligible subjects will sign an informed consent form before any study procedure initiation.

Recording session during hospitalization:

Each subject will undergo up to 15 blood pressure measurement sessions during the hospitalization period. The subject will be connected to the CS6BP device and a cuff simultaneously during the session. There will be at least 30 minutes intervals between the end of the session to the beginning of the next session.

Recording session during follow-up:

The study team personnel may schedule up to 10 follow-up visits with the subject at the clinic or the subject's home for three months following discharge from the hospital. Up to 3 measurement sessions will be conducted during each follow-up visit, maintaining 30 minutes intervals between sessions.

In case of participant discomfort or mechanical hindrance from the watch, the medical staff will stop data collection. The subject can ask to remove the watch during data collection.

ELIGIBILITY:
Inclusion Criteria:

* Age of eighteen (18) year and above
* Ability and willingness to sign an informed consent form

Exclusion Criteria:

* Subjects with hemodynamic support
* Subjects receiving more than 2-3 l of fluid per 24h
* Subjects with septic shock
* Subjects with distal edema
* Subjects with arms trauma, where the watch is not wearable
* Subjects where the radial artery could not be palpate
* Subjects with life expectancy of less than 24h
* Subjects who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the subject's participation in this study
* Any concomitant condition which, in the opinion of the investigator, would not allow safe participation in the study (e.g. drug addiction, alcohol abuse, emotional/psychological diagnosis)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-01-17 (Estimated); Study Completion 2023-01-17 (Estimated)

PRIMARY OUTCOMES:
Performance of CS6BP | up to 1 month
  Assessment of the performance sensitivity of CS6BP in measuring blood pressure
Safety Any adverse event observed during the study will be recorded during the study. | through study completion, an average of 18 months
  Assessment of the safety of using CS6BP for blood pressure measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jacob giris, MD, Principal Investigator — Ichilov Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No